CLINICAL TRIAL: NCT07054424
Title: Development of Repetitive Transcranial Magnetic Stimulation (rTMS) Combined With Machine-assisted Bimanual Therapy (BT) in Upper Limb Rehabilitation
Brief Title: Repetitive Transcranial Magnetic Stimulation Combined With Bimanual Therapy for Upper Limb Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202400379A0C6001
Record Dates: First submitted 2025-06-08; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Post-stroke Upper Limb Hemiparesis; Repetitive Transcranial Magnetic Stimulation (rTMS); Bimanual Therapy; Neuromodulation
Keywords: Stroke; neurorehabilitation; rTMS; bimanual therapy; neuromodulation; upper limb function; theta burst stimulation; brain plasticity
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: An investigator reviewed the inclusion and exclusion criteria and assigned participants to one of the study groups. Participants were randomly allocated to either the rTMS combined with bimanual therapy group, the rTMS only group, or the control group receiving standard rehabilitation. Randomization and group assignment were performed by a research assistant using a computer-generated randomization sequence to ensure unbiased allocation. Each intervention was conducted over a 4-week period, consisting of 10 sessions, during which participants received intervention according to their assigned group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Sham Comparator): 15 mins self-initiated stretching exercise + 50 mins conventional occupational therapy
  Interventions: Other: Conventional occupation therapy; Other: stretching exercise
- rTMS-only group (Active Comparator): 15 mins rTMS and 50 mins conventional occupational therapy
  Interventions: Other: Conventional occupation therapy; Other: rTMS
- rTMS combined with bimanual therapy group (Experimental): 15 mins therapy (rTMS + bimanual therapy) and 50 mins conventional occupational therapy
  Interventions: Other: Conventional occupation therapy; Other: rTMS; Device: bimanual therapy

INTERVENTIONS:
Other: Conventional occupation therapy — Standard occupational therapy focused on improving daily functional skills through task-specific training and adaptive techniques.
Other: stretching exercise — Techniques involving passive or active stretching of muscles to enhance flexibility, reduce spasticity, and prevent contractures.
  Arms: Control group
Other: rTMS — Non-invasive brain stimulation method using magnetic pulses to modulate cortical excitability and promote neural plasticity.
  Arms: rTMS combined with bimanual therapy group; rTMS-only group
Device: bimanual therapy — A training approach that involves simultaneous use of both hands to enhance coordination and functional hand movements through guided exercises, including device-assisted and robot-assisted therapy
  Arms: rTMS combined with bimanual therapy group

SUMMARY:
The goal of this clinical trial is to evaluate whether combining repetitive transcranial magnetic stimulation (rTMS) with machine-assisted bimanual therapy (BT) can improve upper limb function in stroke patients. The participants will be individuals aged 40-80 years who have experienced a first-time ischemic or hemorrhagic stroke. The main questions it aims to answer are:

* Does the combined therapy enhance motor recovery compared to traditional rehabilitation methods?
* Are changes in brain activity associated with improvements in upper limb function?

Participants will be randomly assigned to different groups and will:

* Receive rTMS stimulation on specific areas of the brain to modulate neural activity,
* Perform machine-assisted bimanual exercises to promote motor skills, and
* Undergo assessments before, immediately after, and during follow-up periods to measure functional improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years;
2. First-onset stroke patients;
3. Patients diagnosed with cerebral infarction or hemorrhage through CT or MRI;
4. Signed informed consent form by the patient and their family;
5. Stable physiological parameters;
6. Stroke occurred within the last 12 months;
7. Patients with unilateral hand function impairment caused by the stroke;
8. Upper limb muscle tone (Modified Ashworth Scale, MAS) less than 3 points;
9. Able to follow two-step commands.

Exclusion Criteria:

1. A history of epilepsy or family history of epilepsy;
2. Presence of suicidal tendencies;
3. Currently using medications that lower the seizure threshold;
4. Pregnant or planning to become pregnant;
5. Co-existing neurological diseases (such as multiple sclerosis, other neurodegenerative diseases, meningitis, brain abscess, or meningioma);
6. Subjects with uncontrollable migraines caused by elevated intracranial pressure;
7. Subjects taking antidepressants who cannot discontinue the medication;
8. Subjects with sleep disorders during rTMS treatment;
9. Subjects with cerebellar stroke or brainstem stroke;
10. Cerebral ischemic disorders resulting from traumatic brain injury;
11. Transient ischemic attacks (TIAs);
12. History of bleeding tendency and other conditions affecting upper limb function, such as myasthenia gravis, systemic immune neuropathy, severe epilepsy, endocrine system disorders, wearers of external or internal cardiac pacemakers, individuals with metallic implants or orthopedic devices;
13. Co-existing severe heart, liver, kidney dysfunction, or other serious physical illnesses;
14. Subjects with impaired consciousness who cannot cooperate with examinations or treatments, such as those with mental disorders, or those with intellectual or cognitive impairments, severe dementia;
15. Presence of implanted electronic devices in the body;
16. Co-existing severe liver, kidney, or hematological disorders;
17. Special vulnerable populations;
18. Skin disease (e.g., pressure ulcers, trauma, cellulitis, etc.).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Evaluated at before and after (immediately following the final sessions) the intervention. Additionally, follow-up assessments are conducted at 1 month and 3 months post-treatment to evaluate sustained effects.
  This assessment captures motor recovery across four specific domains: Part A (proximal upper limb-shoulder, elbow, and forearm), Part B (wrist), Part C (hand), and Part D (coordination and speed). The full scale ranges from 0 to 66 and the higher scores represent the better outcome.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Evaluated at before and after (immediately following the final sessions) the intervention. Additionally, follow-up assessments are conducted at 1 month and 3 months post-treatment to evaluate sustained effects.
  This scale is used to evaluate spasticity in muscles by assessing resistance during passive soft-tissue stretching. Scores range from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension), with higher scores indicating greater spasticity.
Upper Extremities Muscle Strength | Evaluated at before and after (immediately following the final sessions) the intervention. Additionally, follow-up assessments are conducted at 1 month and 3 months post-treatment to evaluate sustained effects.
  Manual muscle testing (MMT) is used to assess the strength of major upper limb muscle groups, including the shoulder abductors, elbow flexors/extensors, wrist extensors, and finger flexors/extensors. The scoring is based on the standard 0-5 MMT grading scale, where higher scores indicate greater muscle strength.
Action Reach Arm Test (ARAT) | Evaluated at before and after (immediately following the final sessions) the intervention. Additionally, follow-up assessments are conducted at 1 month and 3 months post-treatment to evaluate sustained effects.
  The ARAT is a standardized observational assessment that evaluates upper limb function through 19 items across four domains: grasp, grip, pinch, and gross movement. The total score ranges from 0 to 57, with higher scores indicating better upper extremity function.
Brunnstrom Recovery Stage | Evaluated at before and after (immediately following the final sessions) the intervention. Additionally, follow-up assessments are conducted at 1 month and 3 months post-treatment to evaluate sustained effects.
  This classification system assesses motor recovery following stroke and categorizes the patient's progress into six stages for the upper extremity, hand, and lower extremity. Stage I represents flaccidity, and Stage VI represents near-normal movement.
Instrumental Activities of Daily Living Scale (IADLs) | Evaluated at before and after (immediately following the final sessions) the intervention. Additionally, follow-up assessments are conducted at 1 month and 3 months post-treatment to evaluate sustained effects.
  The IADLs assess functional independence in more complex daily tasks, including using the telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for own medications, and ability to handle finances. The scores vary by gender: for females, the full 8 items are scored (0-8); for males, traditional scoring omits food preparation, housekeeping, and laundry, resulting in a 5-point scale (0-5). Higher scores indicate greater functional independence.
System Usability Scale (SUS) | Administered once immediately after the final intervention session to capture the participant's impressions of the device's usability.
  The usability of the device and intervention was evaluated using the System Usability Scale (SUS), which captures user experience from both patients and caregivers. The SUS comprises ten Likert-scale items, alternating between positive and negative statements to minimize response bias. Each item is rated from 1 (strongly disagree) to 5 (strongly agree). The total SUS score is calculated and converted to a scale of 0 to 100, with scores above 68 generally indicating acceptable usability.
Satisfaction Questionnaire | Administered once immediately after the final intervention session to assess participants' subjective satisfaction with the intervention.
  A custom satisfaction questionnaire was administered to evaluate participants' overall satisfaction with the rehabilitation process. It uses a 5-point Likert-type scale ranging from 1 (very poor) to 5 (very good) to assess domains such as comfort, perceived effectiveness, motivation, and willingness to continue. Higher scores reflect more favorable responses and higher levels of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, Chang Gung Memorial Hospital at Linkou, Taoyuan 333, Taiwan, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Kim WS, Paik NJ. Safety Review for Clinical Application of Repetitive Transcranial Magnetic Stimulation. Brain Neurorehabil. 2021 Mar 18;14(1):e6. doi: 10.12786/bn.2021.14.e6. eCollection 2021 Mar. PMID 36742107
- [Result] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Result] Liu C, Li L, Li B, Liu Z, Xing W, Zhu K, Jin W, Lin S, Tan W, Ren L, Zhang Q. Efficacy and Safety of Theta Burst Versus Repetitive Transcranial Magnetic Stimulation for the Treatment of Depression: A Meta-Analysis of Randomized Controlled Trials. Neuromodulation. 2024 Jun;27(4):701-710. doi: 10.1016/j.neurom.2023.08.009. Epub 2023 Oct 12. PMID 37831019
- [Result] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Result] Li X, Lin YL, Cunningham DA, Wolf SL, Sakaie K, Conforto AB, Machado AG, Mohan A, O'Laughlin K, Wang X, Widina M, Plow EB. Repetitive Transcranial Magnetic Stimulation of the Contralesional Dorsal Premotor Cortex for Upper Extremity Motor Improvement in Severe Stroke: Study Protocol for a Pilot Randomized Clinical Trial. Cerebrovasc Dis. 2022;51(5):557-564. doi: 10.1159/000521514. Epub 2022 Jan 20. PMID 35051941
- [Result] Chen YM, Lai SS, Pei YC, Hsieh CJ, Chang WH. Development of a Novel Task-oriented Rehabilitation Program using a Bimanual Exoskeleton Robotic Hand. J Vis Exp. 2020 May 20;(159). doi: 10.3791/61057. PMID 32510515
- [Result] Huang JJ, Pei YC, Chen YY, Tseng SS, Hung JW. Bilateral Sensorimotor Cortical Communication Modulated by Multiple Hand Training in Stroke Participants: A Single Training Session Pilot Study. Bioengineering (Basel). 2022 Nov 24;9(12):727. doi: 10.3390/bioengineering9120727. PMID 36550934
- [Result] Chen JL, Ros T, Gruzelier JH. Dynamic changes of ICA-derived EEG functional connectivity in the resting state. Hum Brain Mapp. 2013 Apr;34(4):852-68. doi: 10.1002/hbm.21475. Epub 2012 Feb 17. PMID 22344782
- [Result] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761
- [Result] De Weerdt WJG, Harrison MA. "Measuring recovery of arm-hand function in stroke patients: a comparison of the Brunnstrom-Fugl-Meyer test and the Action Research Arm test. Physiotherapy Canada. 1985; 37:65-70.
- [Result] Crow JL, Lincoln NB, Nouri FM, De Weerdt W. The effectiveness of EMG biofeedback in the treatment of arm function after stroke. Int Disabil Stud. 1989 Oct-Dec;11(4):155-60. doi: 10.3109/03790798909166667. PMID 2701823
- [Result] CARROLL D. A QUANTITATIVE TEST OF UPPER EXTREMITY FUNCTION. J Chronic Dis. 1965 May;18:479-91. doi: 10.1016/0021-9681(65)90030-5. No abstract available. PMID 14293031
- [Result] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Result] Fugl-Meyer AR. Post-stroke hemiplegia assessment of physical properties. Scand J Rehabil Med Suppl. 1980;7:85-93. No abstract available. PMID 6932734
- [Result] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616

DOCUMENTS (1):
  • Study Protocol (2025-04-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT07054424/Prot_000.pdf